CLINICAL TRIAL: NCT00093405
Title: A Phase II Study Of 17-N-Allylamino-17-Demethoxy Geldanamycin (17-AAG)In Metastatic Renal Cell Carcinoma
Brief Title: 17-N-Allylamino-17-Demethoxygeldanamycin in Treating Patients With Metastatic Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000387952; MSKCC-04082; NCI-6479
Record Dates: First submitted 2004-10-06; First posted 2004-10-08 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2005-11

CONDITIONS: Kidney Cancer
Keywords: recurrent renal cell cancer; stage IV renal cell cancer; clear cell renal cell carcinoma
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — tanespimycin

INTERVENTIONS:
Drug: tanespimycin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as 17-N-allylamino-17-demethoxygeldanamycin, work in different ways to stop tumor cells from dividing so they stop growing or die. 17-N-allylamino-17-demethoxygeldanamycin may also stop the growth of tumor cells by blocking the enzymes necessary for their growth.

PURPOSE: This phase II trial is studying how well 17-N-allylamino-17-demethoxygeldanamycin works in treating patients with metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of 17-N-allylamino-17-demethoxygeldanamycin (17-AAG) in patients with metastatic papillary or clear cell renal cell carcinoma.

Secondary

* Determine the safety of this drug in these patients.
* Correlate tumor c-met expression with response in patients treated with this drug.

OUTLINE: This is an open-label study. Patients are stratified according to histology (papillary vs clear cell).

Patients receive 17-N-allylamino-17-demethoxygeldanamycin (17-AAG) IV over 60-90 minutes on days 1, 4, 8, and 11. Treatment repeats every 21 days for up to 1 year in the absence of disease progression or unacceptable toxicity.

Patients are followed at 3 weeks and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 24-74 patients (12-37 per stratum) will be accrued for this study within 6-20 months (clear cell stratum) and 2-5 years (papillary stratum).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed renal cell carcinoma

  * Papillary OR clear cell histology

    * If other histologies are present, clear cell or papillary must be predominant
  * Metastatic disease
* Measurable disease

  * At least 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
* No brain metastases unless previously treated with radiotherapy or surgery AND asymptomatic with no active brain metastases detectable by CT scan or MRI for ≥ 6 months

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 70-100%

Life expectancy

* Not specified

Hematopoietic

* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* AST and ALT ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN

Renal

* Creatinine ≤ 2.0 times ULN

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No severe valvular disease

Pulmonary

* No severe debilitating pulmonary disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No allergy to egg or egg products
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to 17-N-allylamino-17-demethoxygeldanamycin (17-AAG)
* No active or ongoing infection requiring IV antibiotics
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled illness

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No more than 1 prior cytokine-based regimen
* No concurrent biologic therapy

Chemotherapy

* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)

Endocrine therapy

* Not specified

Radiotherapy

* More than 4 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery

* More than 4 weeks since prior major surgery

Other

* Recovered from prior therapy
* No more than 1 prior non-cytokine-based regimen
* No other prior systemic treatment regimens
* No other concurrent cytotoxic therapy
* No other concurrent anticancer therapy
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-08; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Efficacy (complete and partial response)

SECONDARY OUTCOMES:
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Gnanamba V. Kondagunta, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Ronnen EA, Kondagunta GV, Ishill N, Sweeney SM, Deluca JK, Schwartz L, Bacik J, Motzer RJ. A phase II trial of 17-(Allylamino)-17-demethoxygeldanamycin in patients with papillary and clear cell renal cell carcinoma. Invest New Drugs. 2006 Nov;24(6):543-6. doi: 10.1007/s10637-006-9208-z. PMID 16832603